CLINICAL TRIAL: NCT00031759
Title: Phase II Topical Immunomodulatory Therapy With Imiquimod for the Chemoprevention of Recurrent and High-Grade Cervical Intraepithelial Neoplasia (CIN)
Brief Title: Imiquimod in Preventing Cervical Cancer in Women With Cervical Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCCTG-989251; CDR0000069223 (Registry Identifier: PDQ (Physician Data Query)); NCI-P02-0208
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ablative or excisional therapy (Other): Patients undergo ablative or excisional therapy.
  Quality of life is assessed at baseline, 3-5 days after ablation or excisional therapy, at 3 months, and then annually thereafter.
  Patients are followed every 3-4 months until 2 consecutive normal Pap smears or colposcopic exams, every 6 months for 2 years, and then annually until 5 years after completion of study therapy.
  Interventions: Procedure: Ablative or excisional therapy
- Ablative or excisional therapy + imiquimod (Experimental): Patients have topical imiquimod applied to the cervix for 6-10 hours twice weekly for a total of 5 doses. Within 3-4 weeks after the final application, patients undergo ablative or excisional therapy. Quality of life is assessed at baseline, after last dose of study drug, 3-5 days after ablation or excisional therapy, at 3 months, and then annually thereafter.
  Patients are followed every 3-4 months until 2 consecutive normal Pap smears or colposcopic exams, every 6 months for 2 years, and then annually until 5 years after completion of study therapy.
  Interventions: Drug: imiquimod; Procedure: Ablative or excisional therapy

INTERVENTIONS:
Drug: imiquimod
  Arms: Ablative or excisional therapy + imiquimod
Procedure: Ablative or excisional therapy

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain substances to try to prevent the development of cancer. Applying topical imiquimod before abnormal cervical cells are removed may be effective in preventing cervical cancer.

PURPOSE: Randomized phase II trial to study the effectiveness of applying topical imiquimod before abnormal cervical cells are removed in preventing cervical cancer in patients who have recurrent or persistent cervical neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the chemopreventive efficacy of topical imiquimod followed by local ablative or excisional therapy vs ablative/excisional therapy alone in patients with recurrent or high-grade cervical intraepithelial neoplasia.
* Compare the toxicity of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.
* Determine the safety and tolerability of imiquimod in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, disease (primary vs recurrent or persistent), severity of dysplasia (grade I vs grade II vs grade III), current tobacco use (yes vs no), planned surgical procedure (excisional vs laser vs cryotherapy vs other), and time since first abnormal Pap smear, including pathology of ascus favor dysplasia (less than 1 year vs 1-3 years vs more than 3 years). Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo ablative or excisional therapy.
* Arm II: Patients have topical imiquimod applied to the cervix for 6-10 hours twice weekly for a total of 5 doses. Within 3-4 weeks after the final application, patients undergo ablative or excisional therapy.

Quality of life is assessed at baseline, after last dose of study drug (arm II only), 3-5 days after ablation or excisional therapy, at 3 months, and then annually thereafter.

Patients are followed every 3-4 months until 2 consecutive normal Pap smears or colposcopic exams, every 6 months for 2 years, and then annually until 5 years after completion of study therapy.

PROJECTED ACCRUAL: A total of 66-152 (33-76 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary grade II or III cervical intraepithelial neoplasia (CIN) or persistent grade I-III CIN (dysplasia that is not new and requires treatment)
* Squamous cell lesions not involving endocervix by colposcopy OR colposcopy with negative cytobrush or endocervical curettage
* No untreated cervical or vaginal infection other than human papilloma virus
* No desire for hysterectomy as ablative therapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Life expectancy:

* At least 5 years

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* HIV negative
* No AIDS
* No known hypersensitivity to imiquimod
* No latex allergy

PRIOR CONCURRENT THERAPY:

Other:

* No concurrent immunosuppressive therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1999-06; Primary Completion 2004-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 7.5 years

SECONDARY OUTCOMES:
Compare the quality of life of patients treated with these regimens | Up to 7.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bobbie S. Gostout, MD, Study Chair — Mayo Clinic
Locations (8):
- United States (8):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Pachman DR, Barton DL, Clayton AC, McGovern RM, Jefferies JA, Novotny PJ, Sloan JA, Loprinzi CL, Gostout BS. Randomized clinical trial of imiquimod: an adjunct to treating cervical dysplasia. Am J Obstet Gynecol. 2012 Jan;206(1):42.e1-7. doi: 10.1016/j.ajog.2011.06.105. Epub 2011 Jul 13. PMID 21907959